CLINICAL TRIAL: NCT04640961
Title: A Prospective Study of a Single Injection Cross-linked Sodium Hyaluronate Combined With Triamcinolone Hexacetonide (CINGAL®) to Provide Symptomatic Relief of Osteoarthritis of Shoulder Joint
Brief Title: Study of Cingal® for Symptomatic Relief of Osteoarthritis of Shoulder Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cingal 20-02
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Shoulder
Keywords: Sodium Hyaluronate; Triamcinolone Hexacetonide
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cingal (Experimental): Single injection of Cingal into the shoulder joint of subjects diagnosed with osteoarthritis of the shoulder.
  Interventions: Device: Cingal

INTERVENTIONS:
Device: Cingal — Single injection into the shoulder joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH).

SUMMARY:
This Trial will obtain clinical data to support an expanded indication for a single injection of Cingal used for the symptomatic relief of osteoarthritis in the shoulder joint.

DETAILED DESCRIPTION:
Single injection into the shoulder joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH). Participants to be followed to 6 Months post-injection.

ELIGIBILITY:
Screening Inclusion Criteria

1. Age 18 years or older
2. Body Mass Index (BMI) ≤ 35 kg/m2
3. Diagnosis of symptomatic osteoarthritic joint in the index shoulder (Kellgren-Lawrence grade I to III or Guyette grade I to III) to be treated with CINGAL injection.
4. Failed conservative treatment for joint osteoarthritis.
5. NRS pain ≥4 and ≤9 in the index shoulder.
6. Subject must be willing to abstain from other treatments of the index shoulder for the duration of the study.
7. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
8. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up assessment, the subject is willing to discontinue use of acetaminophen/paracetamol.
9. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
10. Able and willing to provide signed informed consent.

Baseline Inclusion Criteria

1. NRS pain ≥4 and ≤9 in index shoulder

Screening Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan or corticosteroids
2. Infection or skin disease in the area of the injection site or index shoulder
3. NRS pain > 3 in the contralateral shoulder
4. Subject received an injection of Hyaluronic Acid (HA) and/or steroid in either joint within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either joint during the course of this study.
5. Known inflammatory or autoimmune disorders (including rheumatoid arthritis, gout), or other pre-existing medical conditions that, in the opinion of the investigator, could impact treatment of the index shoulder or affect the ability of the subject to accurately complete the study questionnaires and comply with the study requirements.
6. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
7. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index shoulder only) corticosteroid within 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index joint is allowed.
8. Significant trauma to the index shoulder within 26 weeks of screening.
9. Chronic use of narcotics or cannabis.

Baseline Exclusion Criteria

1. Subject has a decrease of ≥ 2 in the NRS pain from Screening to Baseline in the index shoulder.
2. Subject has a contraindication to continue with the study treatment injection based on the visual appearance of the synovial fluid aspirate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Anika Therapeutics
Locations (4):
- Krajská zdravotní, a.s. - Masarykova nemocnice Ústí nad Labem, o.z., Ústí nad Labem, Czechia
- Poland (3):
  - NZOZ MEDI-SPATZ M.Spatz, Gliwice
  - SPORTO sp. z o.o, Lodz
  - Przychodnia Rodzinna na Sadowej, Torun

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cingal
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cingal: Single injection into the hip joint of a 4 ml unit dose of Cingal containing 88 mg (22 mg/ml) of cross-linked sodium hyaluronate and 18 mg (4.5 mg/ml) of triamcinolone hexacetonide (TH).
Arm/Group | Cingal
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.12 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Index Shoulder [Count of Participants; unit: Participants]
  Right | 17
  Left | 8

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain
Description: Reduction of Index Shoulder Numerical Rating Scale (NRS) Pain from baseline to 6 months post injection was obtained from participant responses. The NRS Pain Score is an 11-point Likert scale ranged from 0 = No Pain to 10 = Worst Pain level. A negative value for the change in NRS Pain Score indicates less pain post-treatment. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -3.72 (2.19)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

2. Secondary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH) Score
Description: Improvement in pain and function in the index shoulder from baseline to 6 months as measured by the Disabilities of the Arm, Shoulder and Hand (DASH) score. The DASH is a 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores for each question range from 0 (no pain or disability) to 100 (most severe pain or disability) and are averaged to calculate the final DASH score from 0 to 100. A negative value for the change in DASH score indicates improvement. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -38.40 (14.89)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

3. Secondary Outcome: Patient Global Assessment (PGA) Score
Description: The change from baseline to 6 months in index shoulder pain post-treatment as measured by the Patient Global Assessment (PGA) Score. PGA Score records participant responses to their assessment of how much their STUDY (treated) shoulder is bothering them today . The PGA Score is a validated 11-point Likert scale from 0 = No Pain to 10 = Worst Pain.
  A negative value for the change from baseline indicates improvement in PGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cingal
Number analyzed (Participants) | 25
score on a scale | -3.88 (2.35)
Statistical Analysis 1: Comparison: Cingal; Test type: Other; p < 0.0001, ANOVA — P-Value was calculated

4. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. A Calculated Percentage (%) of Participants Responding to Treatment
Description: The post-treatment responder rate is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of participants that met the criteria to be a good responder to treatment. The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better outcome
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 24

5. Secondary Outcome: Usage of Rescue Medication (Acetaminophen/Paracetamol). Number of Participants NOT Using Rescue Medication.
Description: The usage of Rescue Medication (RM) as based on the number of participants at 6 Months post treatmentthat were NOT using acetominophen/paracetamol RM for pain or discomfort.
  A larger percentage of participants that were NOT using RM may correlate to a better clinical outcome in terms of pain.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Cingal
Number analyzed (Participants) | 25
Participants | 21

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the Baseline Study Visit until Study Completion at 26 Weeks.
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Cingal
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=25)
Myocardial Infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cingal (N=25)
Headache (Nervous system disorders) | 3 (3)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Ovulation Pain (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish the Data/Results with the consent of the SPONSOR if:

1. Publication is done after primary publication covering data from all participating sites, and provided the Data/Results do not contain any Confidential Information.
2. Eighteen (18) months has elapsed after entire completion of the Clinical Trial at all participating sites.

DOCUMENTS (2):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04640961/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT04640961/SAP_001.pdf